CLINICAL TRIAL: NCT03681730
Title: A Pragmatic Randomized Controlled Trial of Virtual Reality vs Standard-of-Care for Comfort During Intravenous Catheterization
Brief Title: Virtual Reality vs Standard-of-Care for Comfort During Intravenous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ran Goldman, Professor and Co-head of the Division of Clinical Pharmacology, Division of Emergency Medicine, Department of Pediatrics; Investigator, BC Children's Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-00771
Record Dates: First submitted 2018-07-05; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Intravenous Catheterization
Keywords: Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants are distracted by wearing the virtual reality headset and watching a roller coaster app during an IV start.
  Interventions: Device: Virtual Reality
- Control (Standard-of-Care) (No Intervention): Participants are distracted with Standard-of-Care by doctors, nurses, nurse practitioners, child life specialists and/or parents.

INTERVENTIONS:
Device: Virtual Reality — Participants wear a Virtual Reality headset that consists of a ASUS phone and a VOX+ Z3 3D Virtual Reality Headset. The phone runs the VR Roller Coaster app to produce the virtual environment.
  Arms: Virtual Reality

SUMMARY:
Children often need an intravenous catheter placement for delivery of fluids and medications, a procedure associated with pain and anxiety. In the Emergency Department topical anesthetics are frequently used.

Virtual Reality (VR) is an immersive experience using sight, sound, and position sense. Using VR may enhance distraction during the painful procedure and may reduce attention to pain.

This study will randomize children (6 - 16 years old) to receive Virtual Reality or standard of care in addition to topical anaesthetics during IV placement procedure. Investigators will measure pain, anxiety and satisfaction, amount of analgesics used and the level of success in placing the IV and compare between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 - <17
* The managing physician determines a need for an intravenous catheterization (IV) procedure
* Parents will sign a consent form and children will sign an assent form

Exclusion Criteria:

* Children with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay, autism, others)
* Triage Category 1 (resuscitation)
* Facial features or injury prohibiting wearing the VR goggles

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain using the Faces Pain Scale - Revised. | Pain is reported by children immediately following completion of the IV start
  Level of pain as reported by children using Faces Pain Scale - Revised. The scale includes six faces that represent progressively more intense features of pain. Children point to the face that best represents their current level of pain. The minimum score is 0 (representing least pain) and the maximum score is 10 (representing greater pain). The scale increase in increments of 2.

SECONDARY OUTCOMES:
Anxiety using the Venham Situational Anxiety Score | Anxiety is reported by children immediately following completion of the IV start
  Level of Situational Anxiety as reported by children using the Venham Situational Anxiety Score. This scale includes 8 sets of 2 images of children which represent differing levels of anxiety. Children point to the child that best represents them in that instance. In each set of 2 images of children, one represents greater anxiety (scored as 1) and one represents lesser anxiety (scored as 0). The points from each set of images are totaled. The minimum score is 0 (least anxious) and maximum score is 8 (most anxious).
Patient Satisfaction determined by Global Rating Scale | Satisfaction questions are reported by children immediately following completion of the IV start
  Satisfaction from the procedure is determined by asking 4 questions on a global rating scale. This scale goes from 0-10 where 0 represents "not very much" and 10 represents "very much." Questions are developed from previous virtual reality research. "Overall, how satisfied are you with pain management during plastic surgery?" "Overall, how satisfied are you with anxiety management during plastic surgery?" "To what extent did you feel like you went into the virtual world?" "How much fun did you have while playing in the virtual world?" These questions will be analyzed individually not summed.
Patient Satisfaction determined qualitatively by an open ended question | Satisfaction questions are reported by children immediately following completion of the IV start
  Satisfaction from the procedure is determined qualitatively. Children are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).
Parent Satisfaction determined qualitatively by an open ended question | Satisfaction question is reported by parents immediately following completion of the IV start
  Satisfaction from the procedure is determined qualitatively. Parents are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).
Medication Dose | These will be recorded during the procedure and immediately following the procedure using the patient chart and nursing notes
  How much topical or local anesthetics are used and when they are used (24 hour time); how much sedatives are used and when they are used (24 hour time); how much analgesics are used and when they are used (24 hour time).
Number of IV Trials Until Success | This number will be collected during the procedure
  How many attempts the nurses need to get a functional IV catheter (concealed objective to avoid a Hawthorne effect).
Timing | Documented immediately after patient and family given discharge paperwork
  Time in minutes from readiness for procedure (availability of child, staff and equipment) until completion of procedure (nurse does not need to touch the patient anymore) and until discharged from the emergency department (given discharge paperwork).

CONTACTS AND LOCATIONS:
Overall Officials: Ran D Goldman, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldman RD, Behboudi A. Virtual reality for intravenous placement in the emergency department-a randomized controlled trial. Eur J Pediatr. 2021 Mar;180(3):725-731. doi: 10.1007/s00431-020-03771-9. Epub 2020 Aug 10. PMID 32779029